CLINICAL TRIAL: NCT01670422
Title: Risk Factors Associated With Recurrence and Life-threatening Complications for Patients Hospitalized With Chronic Suppurative Osteomyelitis of the Jaw
Brief Title: Risk Factors Associated With Recurrence and Life-threatening Complications for CSOJ
Status: Completed | Type: Observational
Sponsor: West China College of Stomatology (Other)
Responsible Party: Principal Investigator, Lin Chen, Risk factors associated with recurrence and life-threatening complications for patients hospitalized with chronic suppurative osteomyelitis of the jaw, West China College of Stomatology
Other Study IDs: ABT-1233-RV
Record Dates: First submitted 2012-07-31; First posted 2012-08-22 (Estimated); Last update posted 2012-08-22 (Estimated); Status verified 2012-08

CONDITIONS: Suppurative Osteomyelitis of Jaw; Potential Abnormality of Glucose Tolerance
Keywords: CSOJ; recurrence; life-threatening complications; risk factors
MeSH Terms: conditions — Recurrence

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Clinically, recurrence and life-threatening complications are challenging problems for chronic suppurative osteomyelitis of the jaw. There is no quantitative analysis or report about the causes of or risk factors for the two problems. Doctors identify the causes or risk factors only through clinical experience. The investigators performed a retrospective study of 322 patients with chronic suppurative osteomyelitis of the jaw. The risk factors for the above mentioned two problems were analyzed by logistic regression analysis. The investigators found that some of the patients' general conditions, including age, admission temperature, admission white blood cell count, pre-admission antibiotic administration without consultation, location of the lesion, and general patient condition, were the risk factors. The results indicate that doctors should be mindful of those risk factors and that the management should be more aggressive when the above risk factors are present.

DETAILED DESCRIPTION:
This is a retrospective study of 322 patients hospitalized with CSOJ. The socio-demographic and clinical characteristics were recorded. The risk factors for the above two problems were analyzed by logistic regression analysis. Frequency and percentage were used to indicate descriptive research factors. A univariate logistic regression analysis was performed to calculate the odds ratio (OR) and to identify preliminary risk factors. The preliminary risk factors were further identified by multivariate logistic regression analysis.

ELIGIBILITY:
Inclusion Criteria:

* The diagnosis on admission was made on the basis of the presence of sequestra and laminations of periosteal new bone in the pathological area.
* The other diagnostic criteria is that symptoms such as local pain, pyorrhea, fever, swelling, fistula, neuropalsy, odontoseisis, lymphadenopathy, bromopnea, and trismus pain are unresponsive or insensitive to conservative therapy and simple debridement.

Exclusion Criteria:

* Patients without confirmed evidence of CSOJ and (or) without standard treatment (a combination of antimicrobial therapy and surgery consisting of incision and drainage, debridement or sequestrectomy) were excluded.
* Paget's disease, hypercementosis, fibrous dysplasia, and early stage malignant bone tumor were differentially diagnosed and excluded.

Ages: 1 Month to 83 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with a diagnosis of CSOJ who were admitted to our hospital from 1980 to 2009 were investigated. Ultimately, 322 patients were enrolled in the study of life-threatening complications.Patients were divided into four classes according to their age (years): <6, 6-18, 19-65, >65.
Sampling Method: Non-Probability Sample
Enrollment: 322 (Actual)
Dates: Start 1980-01; Primary Completion 2009-01 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Risk factors associated with recurrence and life-threatening complications for patients hospitalized with chronic suppurative osteomyelitis of the jaw | 30 years
  An age from 6-18 years or > 65 years, pre-admission antibiotic administration, a lesion at the mandibular ramus, concurrent maxillofacial space infection (MSI), and conservation of pathogenic teeth were found to be risk factors for recurrence. An age > 65 years, admission temperature > 39 oC, admission white blood cell (WBC) count >15×109/L, pre-admission antibiotic administration, concurrent MSI, pre-existing diabetes, and respiratory difficulty were found to be risk factors for life-threatening complications.

CONTACTS AND LOCATIONS:
Overall Officials: Lin Chen, DMD, Study Chair — West China Hospital of Stomatology
Locations (1):
- West China Hospital of Stomatology, Chengdu, Sichuan, China

REFERENCES:
- [Derived] Chen L, Li T, Jing W, Tang W, Tian W, Li C, Liu L. Risk factors of recurrence and life-threatening complications for patients hospitalized with chronic suppurative osteomyelitis of the jaw. BMC Infect Dis. 2013 Jul 11;13:313. doi: 10.1186/1471-2334-13-313. PMID 23844897